CLINICAL TRIAL: NCT01916291
Title: Safety and Efficacy of Dinoprostone (Propess) in the Women With Premature Rupture of Membrane or Gestational Age <38
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Propess in PROM or GA<38
Record Dates: First submitted 2013-07-29; First posted 2013-08-05 (Estimated); Last update posted 2020-03-24 (Actual); Status verified 2018-09

CONDITIONS: Induction of Labor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Propess insertion (Experimental)
  Interventions: Drug: Propess insertion group

INTERVENTIONS:
Drug: Propess insertion group

SUMMARY:
Dinoprostone(propess) is commonly used for induction of labor in the pregnant women who has intact membrane after 38weeks of gestational age. The investigators study safety and efficacy of dinoprostone in the pregnant women with premature rupture of membrane or GA<38weeks

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who admitted for induction of labor
* Bishop score <= 6

Exclusion Criteria:

* Contraindication to induction of labor
* Active labor
* Vaginal bleeding, unknown origin
* Hypersensitive to Prostaglandin E
* History of asthma, glaucoma
* Infection (birth canal)
* Placental abruption
* Multiparity(>5)
* Pelvic inflammatory disease
* Heart, lung, kidney disease
* Multiple pregnancy
* Major anomaly
* Fetal distress before induction of labor

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 189 (Actual)
Dates: Start 2013-08-25 (Actual); Primary Completion 2018-08-14 (Actual); Study Completion 2019-04-04 (Actual)

PRIMARY OUTCOMES:
Induction success rate after propess insertion | Day 1 after propess insertion

SECONDARY OUTCOMES:
Concentration of prostaglandinE | at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Joong Shin Park, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Hospital, Seoul
  - Seoul Metropolitan Goverment Seoul National University Boramae Medical Center, Seoul